CLINICAL TRIAL: NCT03321617
Title: Glutamate Reducing Interventions in Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Scott Small, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7459; R61MH112800-01 (NIH)
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Clinical High Risk for Psychosis
MeSH Terms: interventions — pomaglumetad methionil; poly(n-octyl methacrylate); LY 2140023

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, phase 1b, multiple dose trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Identity of medications will be blinded having every subject take an equal number of pills (using identical looking tables of placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- POMA 40mg BID (80mg) (Experimental): Subject will take 40mg pomaglumetad methionil (POMA) twice a day for 14 days.
  Interventions: Drug: Pomaglumetad methionil
- POMA 80mg BID (160 mg) (Experimental): Subject will take 80 mg pomaglumetad methionil (POMA) twice a day for 14 days
  Interventions: Drug: Pomaglumetad methionil
- POMA 120mg BID (240mg) (Experimental): Subject will take 120 mg pomaglumetad methionil (POMA) twice a day for 14 days
  Interventions: Drug: Pomaglumetad methionil
- POMA 160 mg BID (320 mg) (Experimental): Subject will take 160 mg pomaglumetad methionil (POMA) twice a day for 14 days
  Interventions: Drug: Pomaglumetad methionil

INTERVENTIONS:
Drug: Pomaglumetad methionil — metabotropic glutamate 2/3 receptor (mGlu2/3R) agonist
  Other Names: POMA; LY2140023

SUMMARY:
Participants will be administered several doses of pomaglumetad (POMA) (low and high doses) over 14 days to individuals at clinical high risk for developing psychosis and use magnetic resonance imaging (MRI) brain imaging to determine whether these doses of POMA are affecting glutamate levels.

DETAILED DESCRIPTION:
A double-blind, randomized, phase 1b, multiple dose trial of 14 days of treatment with POMA (80 mg, 160 mg, 240 mg, 320 mg) in clinical high risk patients to determine which dose, if any, reduces glutamate and metabolism using MRI techniques. The GO NO-GO decision will be whether or not any dose tested in the R61 phase of the trial decreases left hippocampal CA1 region cerebral blood volume (CBV).

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent
* Currently using a reliable form of birth control

Exclusion Criteria:

* Metal implants in body or a history of metal working
* Lifetime diagnosis of asthmatic symptoms within the past 3 years or known sensitivity to contrast agents
* Lifetime diagnosis of renal failure/disease
* Acute neurological, neuroendocrine, or medical disorder including renal insufficiency (CrCl<40 mL/min/1.73m2)
* Lifetime diagnosis of hypertension or diabetes or seizure disorder
* IQ<70
* Acute risk for suicide and/or violence
* Pregnant lactating
* Current abuse of substances (alcohol, cocaine, stimulants, cannabis, opiates, sedative hypnotics)
* Current use or anticipated need for antipsychotics or mood stabilizers (all antipsychotics, also depakote, lithium, lamotrogine, pregabalin or any med with a mechanism of action like gabapentin), probenecid, selective serotonin reuptake inhibitors, tricyclic antidepressants, and monoamine oxidase inhibitors
* More than one previous gadolinium scan

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Small, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants consented to the protocol and underwent screening procedures but were not randomized (did not receive study medication). Reasons for screen fail:
  1-withdrew consent
  1-unable to undergo scan 3-study was paused due to COVID-19 pandemic
Period: Overall Study
Arm/Group | POMA 40mg BID (80mg) | POMA 80mg BID (160 mg) | POMA 120mg BID (240mg) | POMA 160 mg BID (320 mg)
Started | 3 | 3 | 2 | 3
Completed | 2 | 3 | 2 | 2
Not Completed | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: participants who were randomized (received at least one dose of POMA).
Groups:
- Total: Total of all reporting groups
Arm/Group | POMA 40mg BID (80mg) | POMA 80mg BID (160 mg) | POMA 120mg BID (240mg) | POMA 160 mg BID (320 mg) | Total
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 3 | 11
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2 | 4
  Male | 3 | 1 | 2 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 1 | 3 | 2 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 1 | 5
  White | 2 | 1 | 0 | 1 | 4
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Left Hippocampal CA1 Region Cerebral Blood Volume (CBV) From Baseline to Day 14
Description: Effect of POMA on left CA1 CBV as measured by percent change from baseline scan (Time 1) to Day 14 scan (Time 2)
Time Frame: Baseline to 14 days of POMA/placebo
Population: participants who completed both baseline and Day 14 scans
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | POMA 40mg BID (80mg) | POMA 80mg BID (160 mg) | POMA 120mg BID (240mg) | POMA 160 mg BID (320 mg)
Number analyzed (Participants) | 2 | 3 | 2 | 2
Percent change | 0.40684405 (.63605395) | -0.081559 (0.1522939) | 0.0219668 (0.1484273) | -0.0269017 (0)

ADVERSE EVENTS:
Time Frame: From consent to 30 days after last dose of study medication, up to 74 days (30-day screening period, 14-day randomization period, 30 day follow up)
Arm/Group | POMA 40mg BID (80mg) | POMA 80mg BID (160 mg) | POMA 120mg BID (240mg) | POMA 160 mg BID (320 mg)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 1/2 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POMA 40mg BID (80mg) (N=3) | POMA 80mg BID (160 mg) (N=3) | POMA 120mg BID (240mg) (N=2) | POMA 160 mg BID (320 mg) (N=3)
nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
itching/restlessness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT03321617/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT03321617/SAP_001.pdf
  • Informed Consent Form (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT03321617/ICF_002.pdf